CLINICAL TRIAL: NCT02444832
Title: Multicenter Retrospective Registry of Anterior Communicating Artery Aneurysms With Endovascular Therapy
Acronym: MACAARET
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospital Clinic of Barcelona (Other)
Collaborators: Hospitales Universitarios Virgen del Rocío (Other); Hospital Universitario Reina Sofia de Cordoba (Other Government)
Responsible Party: Principal Investigator, Federico Zarco, Neurorradiologist,, Hospital Clinic of Barcelona
Other Study IDs: NeurovascCDI001
Record Dates: First submitted 2015-05-12; First posted 2015-05-15 (Estimated); Last update posted 2015-05-15 (Estimated); Status verified 2015-05

CONDITIONS: Intracranial Aneurysm; Anterior Communicating Artery Aneurysm; Cerebral Aneurysm; Aneurysm, Ruptured
MeSH Terms: conditions — Intracranial Aneurysm; Aneurysm, Ruptured

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Based on the anatomical features of the anterior Communicating artery complex, the investigators will analyze the outcome of the ACoA aneurysms treated by endovascular therapy.

The most common site of intracranial aneurysms is the anterior communicating artery (AcomA). AcomA aneurysms account for approximately one-fourth of all intracranial aneurysms.

Recent publications have addressed specifically the endovascular treatment of AcoA aneurysms. Furthermore, detailed anatomic characteristics and the effects of the multiple variations of the anterior communicating artery complex have scarcely been reported.

The hemodynamic factors play a fundamental role in the adequate treatment of aneurismal coiling.

The objective of our registry is to analyze the impact of morphological configuration of the anterior communicating artery complex and the results of coil embolization in AcoA aneurysms

ELIGIBILITY:
Inclusion Criteria:

* Patient with Anterior Communicating Artery Aneurysm treated with endovascular coiling.

Exclusion Criteria:

* Patients without imaging follow up of at least 12 months after endovascular treatment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Communicating Artery Aneurysm treated with endovascular coiling.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2015-05; Primary Completion 2017-06 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Effective Aneurysm Coiling (no residual cerebral aneurysm) | 1 year

SECONDARY OUTCOMES:
All Cause Mortality | 1 year
Neurological Outcome (classified with the Glasgow Outcome Scale, Rankin Scale) | 1 year
  All patients will be classified with the Glasgow Outcome Scale, Rankin Scale.
Procedural device-related serious adverse events | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Federico Zarco, MD, Principal Investigator — Hospital Clinic of Barcelona
Locations (1):
- Hospital Clinic, Barcelona, Barcelona, Spain

REFERENCES:
- [Background] Elias T, Ogungbo B, Connolly D, Gregson B, Mendelow AD, Gholkar A. Endovascular treatment of anterior communicating artery aneurysms: results of clinical and radiological outcome in Newcastle. Br J Neurosurg. 2003 Jun;17(3):278-86. doi: 10.1080/0268869031000153251. PMID 14565533
- [Background] Moret J, Pierot L, Boulin A, Castaings L, Rey A. Endovascular treatment of anterior communicating artery aneurysms using Guglielmi detachable coils. Neuroradiology. 1996 Nov;38(8):800-5. doi: 10.1007/s002340050352. PMID 8957810
- [Background] Birknes JK, Hwang SK, Pandey AS, Cockroft K, Dyer AM, Benitez RP, Veznedaroglu E, Rosenwasser RH. Feasibility and limitations of endovascular coil embolization of anterior communicating artery aneurysms: morphological considerations. Neurosurgery. 2006 Jul;59(1):43-52; discussion 43-52. doi: 10.1227/01.NEU.0000219220.25721.B9. PMID 16823299
- [Background] Molyneux AJ, Kerr RS, Yu LM, Clarke M, Sneade M, Yarnold JA, Sandercock P; International Subarachnoid Aneurysm Trial (ISAT) Collaborative Group. International subarachnoid aneurysm trial (ISAT) of neurosurgical clipping versus endovascular coiling in 2143 patients with ruptured intracranial aneurysms: a randomised comparison of effects on survival, dependency, seizures, rebleeding, subgroups, and aneurysm occlusion. Lancet. 2005 Sep 3-9;366(9488):809-17. doi: 10.1016/S0140-6736(05)67214-5. PMID 16139655